CLINICAL TRIAL: NCT05195346
Title: A Cross-sectional Survey of HIV Healthcare Providers and People Living With HIV in Thailand, and Their Awareness, Knowledge, and Implementation of Undetectable = Untransmissible
Brief Title: Undetectable = Untransmissible in Thailand (888/64)
Acronym: 888/64
Status: Completed | Type: Observational
Sponsor: Institute of HIV Research and Innovation Foundation, Thailand (Other)
Responsible Party: Sponsor
Other Study IDs: IHRI012
Record Dates: First submitted 2021-12-11; First posted 2022-01-18 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2023-01

CONDITIONS: HIV
Keywords: Undetectable = Untransmissible; Knowledge; Awareness; Implementation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- People Living with HIV (PLHIV): Thai people living with HIV, aged 18 or above, who are on Antiretroviral Therapy (ART)
- HIV Healthcare Providers: Thai healthcare providers, including but not limited to doctors, nurses, counsellors, lay providers, pharmacists, lab technicians, etc., who take care of any persons living with HIV. All aged 18 or above

SUMMARY:
This is a cross-sectional study to assess awareness, knowledge, and implementation of the concept of U=U among Thai PLHIV and Thai HIV healthcare providers, as well as associated factors. Data will be collected on an online survey platform called Alchemer. Questions on the survey will evaluate awareness, knowledge, and implementation of U=U among participants, as well as collect sociodemographic information of participants.

DETAILED DESCRIPTION:
Recruitment

Recruitment will start with the distribution of a brief description of the survey, along with the link to the questionnaire itself. This will be distributed systematically through the use of the snowball sampling method on popular social networking platforms (such as Line, Instagram, WhatsApp, Facebook and Twitter), where 'seed' distributors, who may be categorised into different groups (such as age, gender identity and treatment facility for PLHIV or healthcare facility and type of healthcare provider for HIV healthcare providers), will share out links to a number of friends. Participants will be enrolled into the study once they click on the link leading them to the survey and complete the questionnaire.

Informed consent process

Consent will be obtained by action. A brief description of the survey will be distributed, along with the online link to the survey, which will be on SurveyGizmo. All data will be collected anonymously. A digitalised consent form will be presented to participants before they start the survey, which will outline the potential risks and benefits. All participants will be equal to or over the age of 18; therefore, parental consent is not needed.

Questionnaires

The questionnaire should take no more than 15 minutes to complete. The survey will be completed on Alchemer (formerly SurveyGizmo), a flexible, cross platform online survey software, or other popular online survey platforms with similar features, with the participant giving consent through action. Questions on the survey will evaluate awareness, knowledge, and implementation of U=U among participants, as well as collect sociodemographic information of participants. All the information collected will be kept confidential and anonymous, and participants cannot be identified in any way. There will be two different questionnaires, one for PLHIV and one for HIV healthcare providers; each survey will be slightly altered to for the appropriate participant category. After the questionnaire is completed, participants can choose to be redirected to educational webpages with more information on U=U.

Data analysis

Data used for analysis will only include data that is submitted through the online portal. It will be analysed using descriptive statistics including percentage, mean and standard deviations, as well as inferential statistics such as Chi Square test or t-test depending on the characteristics of data

ELIGIBILITY:
Inclusion Criteria:

1. Thai HIV healthcare providers or Thai PLHIV on ART medication
2. ≥ 18 years of age
3. Can read, understand, and write Thai
4. Provide consent to participate in the study

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will include any HIV healthcare providers or Thai people living with HIV on antiretroviral therapy. All participants must be of Thai nationality and 18 or above years of age.
Sampling Method: Non-Probability Sample
Enrollment: 770 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
To study awareness, knowledge, and implementation of U=U concept among Thai HIV healthcare providers | 12 months
  Questions on the survey will evaluate awareness, knowledge, and implementation of U=U among participants. All the information collected will be kept confidential and anonymous, and participants cannot be identified in any way. Data used for analysis will only include data that is submitted through the online portal. It will be analysed using descriptive statistics including percentage, mean and standard deviations, as well as inferential statistics such as Chi Square test or t-test depending on the characteristics of data. We hypothesised that awareness will be low among Thai HIV healthcare providers (<50%), and thereby knowledge and implementation will be equal to or lower.
To study awareness, knowledge, and implementation of U=U and its physical, mental, and sexual health impacts on Thai PLHIV. | 12 months
  Questions on the survey will evaluate awareness, knowledge, and implementation of U=U among participants. All the information collected will be kept confidential and anonymous, and participants cannot be identified in any way. Data used for analysis will only include data that is submitted through the online portal. It will be analysed using descriptive statistics including percentage, mean and standard deviations, as well as inferential statistics such as Chi Square test or t-test depending on the characteristics of data. We hypothesised that awareness will be relatively low among Thai PLHIV (~50%); therefore, knowledge and implementation will be equal to or lower.
To explore factors associated with awareness, knowledge, and implementation of U=U concept among Thai HIV healthcare providers and Thai PLHIV. | 12 months
  Questions on the survey will also collect sociodemographic information of participants. All the information collected will be kept confidential and anonymous, and participants cannot be identified in any way. Data used for analysis will only include data that is submitted through the online portal. It will be analysed using descriptive statistics including percentage, mean and standard deviations, as well as inferential statistics such as Chi Square test or t-test depending on the characteristics of data. We hypothesised that factors most closely relative to awareness, knowledge, and implementation of U=U among PLHIV could be duration on ART, size of treatment facility, age, and gender identity. Among HIV healthcare providers, likely factors of influence will be size of healthcare facility and type of healthcare provider.

CONTACTS AND LOCATIONS:
Overall Officials: Nittaya Phanuphak, MD,Ph.D, Principal Investigator — INSTITUTE OF HIV RESEARCH AND INNOVATION FOUNDATION
Locations (1):
- Institute of HIV Research and Innovation, Pathum Wan, Bangkok, Thailand